CLINICAL TRIAL: NCT03604952
Title: Effects of Ramadan Observance on Pulmonary Variables, Exercise Performance and Postural Balance in Male Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Ramadan Observance in Male Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Marwa Mekki, Avenue Mohamed Karoui, 4002, Sousse, Tunisia, Faculty of Medicine, Sousse
Other Study IDs: Faculty of Medicine of Sousse,
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease; Ramadan observance; pulmonary variables; postural balance; exercise performance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COPD patients — Tests performed one week before Ramadan (C), and during the second (R-2) and the fourth weeks of Ramadan (R-4)

SUMMARY:
Purpose: To analyze the effects of Ramadan observance (RO) on pulmonary variables, exercise performance and postural balance in patients with chronic obstructive pulmonary disease (COPD).

Methods: Twenty COPD patients (age=72.7 ± 4.1 yr, non-smokers, without cardiac or neuromuscular complications) were evaluated. Tests performed one week before Ramadan (C), and during the second (R-2) and the fourth weeks of Ramadan (R-4) included standard spirometry, a quality of life questionnaire (VQ11), a 6-min walking test (6MWT), measurement of maximal voluntary contraction force of the quadriceps (MVC), Timed Get Up and Go (TUG), Berg Balance Scale (BBS) and Unipedal Stance (UST).

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide ; prevalence is high in Tunisia, with 7.8 % and 4.2 % of the population in disease stages 1 and 2 respectively . Patients with COPD show an impaired exercise tolerance, often with severe dyspnea, a decreased ability to participate in the activities of daily living, and a poor health-related quality of life.

The common practice of those observing Ramadan is to have two meals per day: a large meal shortly after sunset and a much lighter one immediately before dawn. Ramadan observance (RO) is characterized by many changes in diet and sleep patterns , often with a decrease in the time available for nocturnal sleep . Studies in athletes have shown altered muscle metabolism , hormonal changes , and an impaired physical performance depending on the time of day at which test sessions were performed . Sometimes there are disturbances of cognitive function , and Patel et al noted decreases in postural control even in young adults, due to momentary lapses of attention after sleep deprivation . Such changes are of particular concern in elderly patients with COPD, since their ability to carry out the activities of daily living may initially be marginal, and any disturbances of balance and cognitive function associated with RO could increase the risk of falls .

To date, only one previous study has examined the effects of Ramadan observance in patients with COPD ; this report focused almost exclusively upon changes in medication use during RO. Most Muslim patients with COPD observe Ramadan (for example, 93% in Turkey ), but little is known about the clinical and physiological effects of such fasting in COPD .Thus, the aim of the present study was to analyze the effects of RO on pulmonary variables, exercise performance and postural balance in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:Clinically stable individuals with a functional diagnosis of COPD according to the global strategy for the diagnosis, management and prevention of COPD guideline were selected

* medication remained unchanged during Ramadan).Smokers

Exclusion Criteria:

* those with cardiovascular or neurological disease, lower extremity musculoskeletal problems and visual deficits that could affect postural control were excluded

Ages: 67 Years to 77 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants in this study were 20 male volunteers with COPD
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2015-07-14 (Actual); Study Completion 2015-07-16 (Actual)

PRIMARY OUTCOMES:
standard spirometry | 15 MIN
  Pulmonary function was tested using a Zan 100 spirometer (Inspire Health GmbH, Germany) according to Respiratory Society recommendations, with data related to Tunisian norms
6-min walking test | 6 min
  Exercise Performance was assessed by 6MWT , performed indoors, along a flat, straight, 30 m walking course with a tiled surface; chairs were placed in case participants needed to rest
The timed get up and go (TUG), | 15 seconds
  The TUG score reflects both balance and functional mobility . The time taken to stand from a chair, walk a distance of 3 meters, turn around, return to the chair, and sit down was recorded
the Berg balance scale | 10 MIN
  The BBS is a psychometrically robust clinical measurement of balance for older adults. It assesses performance on 5 levels, from 0 (cannot perform) to 4 (normal performance), with14 items involving functional balance control, including transfer, turning and stepping; a perfect score is 56
the Unipedal stance | 45 secondes
  The UST measures the participant's ability to stand on his preferred leg. A unipedal stance is maintained for a long as possible; failure is defined as shifting the stance foot or placing the lifted foot on the floor. The UST was considered normal if the unipedal stance was maintained for 45 seconds or longer

SECONDARY OUTCOMES:
Isometric leg force assessment | 5 secondes
  After a warm-up phase of the leg extensor muscle consisting of 5 min cycling at 60% of maximum HR reached at the end of 6MWT, 3 maximal voluntary isometric contractions (MVC) were made, separated by 5 min rest intervals
Quality of life questionnaire (VQ 11) | 10 min
  The VQ11 is a reliable and valid measure of COPD-specific health related quality of life (HRQoL) [27]. The 11 items cover three main components: functional (dyspnea, fatigue and mobility), psychological (physical confidence, anxiety, depression and sleep), and social (life project, social life, closeness and emotional life). A high total score indicates a poor HRQoL

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Sousse, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No